CLINICAL TRIAL: NCT07213739
Title: A Laboratory Trial to Investigate the Biomechanical and Physiological Responses to Prolonged Lying Postures During CLP When Combined With Pulsation Therapy on Caylis Pro® Low Air Loss (LAL) System
Brief Title: A Trial to Investigate the New Caulis Pro® Low Air Loss (LAL) System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arjo AB (Industry)
Responsible Party: Principal Investigator, Karin Hannander, RN, Director, Arjo AB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CaylisPro-MACC-004-2025
Record Dates: First submitted 2025-09-03; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Health Adult Subjects; Pressure Injury Prevention
Keywords: caylis, Arjo

STUDY DESIGN:
Intervention Model Description: During the test each volunteer will adopt three distinct postures namely supine, lateral lying (pelvis titled to 30°) and cardiac high sitting (head of bed at 45°), while a series of measurements will be performed at the individual-support surface interface.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 study 2 separate session (Other): The healthy volunteers will be placed on a new mattress which has continuous low pressure (CLP and a pulsatio feature) and during that time period different measurements will be taken.
  Interventions: Device: CLP and pulsation

INTERVENTIONS:
Device: CLP and pulsation — As an alternative to manual repositioning, advanced air mattress systems have been introduced to periodically relieve support pressures.
  A number of measurements have been used to examine the performance of support surfaces. As an example, interface pressure measurements between the individual and the support surface have been extensively used in both lab-based and clinical studies . We are now investigation the functions to reduce pressure in our new Caylis mattress

SUMMARY:
Investigation of biomechanical and physiological functions of laying on a new mattress in healthy volunteers.

DETAILED DESCRIPTION:
This trial primary aims to investigate the biomechanical (interface pressure) and physiological (microvascular function) responses to prolonged lying postures during CLP when combined with pulsation therapy on a product not yet placed on the market (Caylis Pro® LAL System).

A secondary aim is to compare the frequency and amplitude of different pulsation modes with respect to the biomechanical and physiological responses at the participant-support surface interface.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Healthy male or female

Exclusion Criteria:

* Systemic skin disease
* History of pressure ulcers in the sacrum or heels
* Diabetes
* Long term steroid use
* Inability to maintain lying posture for prolonged periods

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
This trial primary aims to investigate the biomechanical (interface pressure) and physiological (microvascular function) responses to prolonged lying postures during CLP when combined with pulsation therapy on a product not yet placed on the market. | Day 1 and 2
  * Comfort, support and firmness scores (using a 7 point verbal rating scale )
  * Interface pressure distribution (ForeSitePT, XSensor)
  * Transcutaneous gas levels
  * Microclimate measures between the participant and the support surface using temperature and humidity sensors (Sensiron SH75).
  * Internal Mattress air pressures

IPD SHARING:
Plan to Share IPD: No
This is a single centre study